CLINICAL TRIAL: NCT06606574
Title: PREDICT-ITB: Predicting Response in Children With Dystonic Cerebral Palsy to Intrathecal Baclofen
Brief Title: Intrathecal Baclofen and Pediatric Dystonia
Acronym: PREDICT-ITB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sruthi P. Thomas, MD, PhD, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-54449; R01HD112563 (NIH)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Dystonic Cerebral Palsy
Keywords: Intrathecal baclofen; Spasticity; Dystonia; Cerebral Palsy
MeSH Terms: conditions — Muscle Spasticity; Dystonia; Cerebral Palsy

STUDY DESIGN:
Masking Description: Therapists completing the assessments will be blinded to the patient's baseline characteristics, imaging findings, and current ITB dosage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Titration protocol (Other): This is a single arm study where each subject will be started with a standardized ITB protocol. The dosing will be increased or decreased stepwise based on parameters that have been described in detail in the intervention section.
  Interventions: Other: Titration protocol

INTERVENTIONS:
Other: Titration protocol — A standardized titration protocol for ITB will be used and the ITB dose will be increased to the next step if 1) there is persistent hypertonia identified on the dystonia screener or ASAS total spasticity, or 2) there is room for improvement on the D-FIS, and 3) there are no detrimental side effects (e.g., worsening head control). This will be continued until 1) dystonia and spasticity have been eliminated or no longer deemed as functionally impairing by the medical team, 2) side effects prevent further titration, or 3) a maximum dose of 2000 mcg/day has been reached. Once steady state is reached, this new dose becomes the maintenance dose for the rest of the trial. If there are detrimental side effects, the child will be seen weekly to confirm resolution of side effects. If side effects persist, the child will be reduced at each visit to the previous step. Once side effects are controlled, this new dose becomes the child's maintenance dose for the rest of the trial.

SUMMARY:
The goal of this clinical trial is to better understand the effects of intrathecal baclofen (ITB) on children with dystonic cerebral palsy (CP).

The main questions this study aims to answer are:

(1) Determine if ITB reduces dystonia while identifying other potential benefits, (2) Identify the characteristics of children with the best response to ITB (3) Develop a holistically representative composite outcome measure for dystonic CP.

This study will evaluate patient improvement by using a standardized titration, or medication management, protocol to gradually increase the childs ITB dosages over a 12-month period until they achieve maximum benefit with minimal to no side effects. This titration protocol mimics what is currently done through routine care but with more precision. This study will also directly measure the global effects of ITB, taking into account spasticity, known dystonia triggers (e.g. pain), and patterns of CNS injury that cause dystonia.

Participants will:

1. Complete a total of 4 additional clinic visits outside usual care. These appointments will be with physical and occupational therapists as well as the study PI to complete evaluations for dystonia, spasticity, and function.
2. Complete several questionnaires at these visits. The total duration of the study for an individual child will be 12 months.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of physical disability in childhood and affects ~1 in 323 in the US per the CDC. The lifetime medical costs for an individual with CP was expected to be ~$1.4 million (inflation adjusted). An effective way to improve quality of life and decrease disease burden, both in childhood and adulthood, is to significantly reduce or eliminate abnormal tone. As muscle tone subsides, it is easier to move the body both passively and actively. A reduction in tone can improve quality of life, reduce pain, ease the burden of daily care and performance of day-to-day activities, and reduce healthcare costs. Intrathecal baclofen ( ITB) is used widely to manage dystonia in CP even though the data on exact efficacy is mixed. Therefore, the goal of this study, is to understand the effects of ITB on a heterogenous population of children with dystonic CP.

The goal of the proposed research is to complete a longitudinal prospective cohort study investigating the effects of intrathecal baclofen (ITB) on children with dystonic cerebral palsy (CP). This study builds on new preliminary data and capitalizes on the expertise of an established transdisciplinary team, a high-resource academic clinical environment, and a diverse Parent-Patient Council. The study's findings are likely to have high impact to improve future treatment of children with dystonic CP, including identifying key patient characteristics associated with more or less positive outcomes and developing a sensitive, efficient multidimensional composite measure to assess treatment responsiveness. Specifically, this protocol aims to determine the 12-month effects of ITB in a cohort of 65 clinically representative, ITB naïve, children with dystonic CP using a standardized titration protocol. Additionally, this protocol aims to complete a detailed characterization of brain malformation and injury patterns in children with dystonic CP and explore potential differences in outcome patterns as related to patient characteristics and use findings to guide development of a sensitive multidimensional or composite measure that captures clinically important areas of change for the child and family.

Our study site will be Texas Children's Hospital (TCH) in Houston, TX, our PI Sruthi Thomas' home institution. TCH has over 860 active patients with CP and just over 200 patients with ITB. Houston, TX, is the most diverse city in the United States, allowing us to recruit a very diverse patient population based on ethnicity and socioeconomic groups.

ELIGIBILITY:
Inclusion Criteria:

* Child must be large enough to have an ITB pump implanted (typically ~18 kg/4 years old)
* They have a diagnosis of CP
* Presence of dystonia verified with a documented Hypertonia Assessment Tool (HAT) and they must have a Barry-Albright Dystonia Scale (BADS) score >15
* They have been identified by a physician for ITB treatment for tone management and the family/child have agreed to proceed with implantation; note: an ITB trial dose is not necessary to qualify
* Child and family are willing to participate in full schedule of formal assessments, spanning pre-implantation, every 2 weeks until ideal intrathecal baclofen pump dosing is reached, and follow-up assessments

Exclusion Criteria:

* Emergent need for ITB such as status dystonicus or paroxysmal sympathetic hyperactivity
* Botulinum injections within 3 months or phenol injections within 6 months of enrollment
* Foster care placement or incarceration

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Barry-Albright Dystonia Scale (BADS) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The BADS was created based on the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS), a tool originally designed to detect cervical dystonia in adults.The BADS tailors this scale for detecting dystonia in CP and acquired brain injury in individuals with limitations in cognition and physical ability. Scoring focuses on posturing and involuntary dystonic movements to detect potential changes in dystonia that affect ease of care and comfort. It does not assess functional tasks. It has moderate internal consistency and inter-rater reliability. It has effectively detected change with ITB. The BADS was also found to have the greatest clinical utility for children with dystonic CP

SECONDARY OUTCOMES:
Dyskinesia Impairment Scale-II (DIS-II) | Baseline (pre-ITB initiation), 3 months, 6 months, 12 months post ITB initiation
  The DIS-II is one of the newest scales to measure dystonia and choreoathetosis at rest and during activity. It is unique in separating choreoathetosis from dystonia in this population. It has moderate internal consistency and fair interrater reliability. We include this measure because it was a key measure in the IDYS trial by Bonouvrie LA et al., the single RCT trial, thus permitting direct comparison across our studies.
Australian Spasticity Assessment Scale (ASAS) and Composite Measure | Baseline (pre-ITB initiation), 3 months, 6 months, 12 months post ITB initiation
  The ASAS combines the best aspects of the MTS with the simplicity of the MAS's scoring system. It has clear instructions on how the limb must be tested while supine to increase reproducibility. Its interrater reliability is very high with a weighted kappa of 0.87, making it ideal for a large study with multiple time points. We will generate a composite score (as well have individual scores) for key muscle groups.
Modified Ashworth Scale (MAS) | Baseline (pre-ITB initiation), 3 months, 6 months, 12 months post ITB initiation
  While our study relies strongly on the ASAS, we will also measure MAS so our data can be compared across studies.
Gross Motor Function Measure (GMFM) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The GMFM is an assessment tool to measure changes in gross motor function with interventions in children with CP. Given that children enrolled in this study will fall in the GMFCS IV-V category, we will not score section E: walking, running, and jumping. As a widely used clinical and research tool, it has an excellent test-retest reliability and excellent inter- and intrarater reliability. The minimal clinically important difference (MCID) is ~0.7-1.2 points in ambulatory children with CP but unfortunately a level has not been determined for non-ambulatory children.
Box and Blocks Test | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  This test is a quick, simple way to assess manual dexterity. This test cannot be used in a child with severe upper extremity impairment or severe cognitive impairment, therefore, not all participants in this study will be able to complete this task. A child is asked to move as many blocks as possible from one side of a divided box to the other in 60 seconds. It has excellent interrater reliability and MCID of 5.29- 6.46 seconds.
Performance Quality Rating Scale (PQRS) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The PQRS is an observational measure of performance quality of a parent/patient-selected meaningful activity. Occupational therapists use a video recording of a child performing the task of interest and then rate the quality. It has high interrater reliability from 0.83-0.93 and test-retest reliability >0.80.
Canadian Occupational Performance Measure (COPM) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The COPM focuses on occupational performance in all areas of life, including self-care, leisure, and productivity. It consists of a semi- structured interview to determine areas of concern for the parent and child. Together with an occupational therapist, they score performance on the particular concerns at the set timepoints in the study. We will have families and children set 2-3 goals that are relevant to ITB treatment. The COPM is an excellent tool for this study as it is very sensitive to change and has an established MCID of 2 points.
Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD©) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The CPCHILD© measures a child with severe disability's overall health, comfort, function, and QoL in relationship to their medical conditions. It has 37 questions answered by the child or parent about activities of daily living, positioning, transferring and mobility, comfort and emotions, communications and social interaction, health, and overall QoL. It was initially validated in children with CP and traumatic brain injuries. Prospective longitudinal cohort studies are underway to assess the measure's responsiveness/sensitivity to change.
Patient-Reported Outcomes Measurement Information System (PROMIS®) Questionnaires | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  NIH's Office of Strategic Coordination - Common Fund's PROMIS® developed a validated item bank of patient-reported outcomes for clinical research and practice. The PROMIS offers many short form questionnaires that are simple and quick for parents and children to complete. We will use the following to assess pain, anxiety, depression, and stress:
  (1a) PROMIS® Pediatric Item Bank v1.0 - Pain Behavior 8a
  (1b) PROMIS® Parent Proxy Bank v1.0 - Pain Behavior 8a. (2a) PROMIS® Pediatric Item Bank v2.0 - Pediatric Anxiety - Short Form 8a (2b) Parent Proxy Bank v2.0 - Parent Proxy Anxiety - Short Form 8a (3a) PROMIS® Pediatric Item Bank v2.0 - Pediatric Depressive Symptoms - Short Form 8a (3b) Parent Proxy Bank v2.0 - Parent Proxy Depressive Symptoms - Short Form 6a. (4) PROMIS® Parent Proxy Bank v1.0 - Psychological Stress Experiences - Short Form 4a.
  (5) PROMIS® Parent Proxy Bank v1.0 - Physical Stress
Goal Attainment Scale (GAS) | Baseline (pre-ITB initiation) , 3 months, 6 months, 12 months post ITB initiation
  The GAS is a unique outcome measurement tool with some controversy about its standardization. It selects a single important goal to be tracked before, during, and after an intervention. GAS was created to account for the heterogeneity of the rehabilitation population. In addition to choosing the goal(s), the child and their family, with guidance from their care team, choose how to define a successful outcome. GAS is tailored to each child and has been shown to be as sensitive to change over time as other standard outcome measurement tools, including the GMFM (discussed above) and the Pediatric Evaluation of Disability Inventory. The single RCT IDYS trial used the GAS as their 1o outcome measure. By including this, we can directly compare results.

CONTACTS AND LOCATIONS:
Overall Officials: Sruthi P Thomas, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Childrens Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant data and final study results may be reviewed with the participant(s) and their families. Data de-identified data may be summarized into graphs showing the changes in all of the measures at 0, 3, 6, and 12 months.

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Economic costs associated with mental retardation, cerebral palsy, hearing loss, and vision impairment--United States, 2003. MMWR Morb Mortal Wkly Rep. 2004 Jan 30;53(3):57-9. PMID 14749614
- [Background] Lungu C, Ozelius L, Standaert D, Hallett M, Sieber BA, Swanson-Fisher C, Berman BD, Calakos N, Moore JC, Perlmutter JS, Pirio Richardson SE, Saunders-Pullman R, Scheinfeldt L, Sharma N, Sillitoe R, Simonyan K, Starr PA, Taylor A, Vitek J; participants and organizers of the NINDS Workshop on Research Priorities in Dystonia. Defining research priorities in dystonia. Neurology. 2020 Mar 24;94(12):526-537. doi: 10.1212/WNL.0000000000009140. Epub 2020 Feb 25. PMID 32098856
- [Background] Bohn E, Goren K, Switzer L, Falck-Ytter Y, Fehlings D. Pharmacological and neurosurgical interventions for individuals with cerebral palsy and dystonia: a systematic review update and meta-analysis. Dev Med Child Neurol. 2021 Sep;63(9):1038-1050. doi: 10.1111/dmcn.14874. Epub 2021 Mar 27. PMID 33772789
- [Background] Bonouvrie LA, Becher JG, Vles JSH, Vermeulen RJ, Buizer AI; IDYS Study Group. The Effect of Intrathecal Baclofen in Dyskinetic Cerebral Palsy: The IDYS Trial. Ann Neurol. 2019 Jul;86(1):79-90. doi: 10.1002/ana.25498. Epub 2019 May 21. PMID 31050023
- [Derived] Thomas SP, Fehlings D, Ramey S, Conaway M, Kralik S, Raskin J. PREDICT-ITB: Predicting response in children with dystonic CP to ITB - study protocol. medRxiv [Preprint]. 2025 Jul 8:2025.07.08.25331080. doi: 10.1101/2025.07.08.25331080. PMID 40672491